CLINICAL TRIAL: NCT06469892
Title: Application of Salivary and Plasma Exosomes in the Diagnosis of Oral Leukoplakia Malignant Transformation and Prognosis Monitoring of Oral Cancer
Brief Title: Saliva and Plasma Exosomes for Oral Leukoplakia Malignant Transformation Diagnosis and Oral Cancer Prognosis Monitoring
Status: Completed | Type: Observational
Sponsor: Beijing Stomatological Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaobing Guan, Doctor and Professor of Oral Medicine，and Director of Department of Oral Medicine, Beijing Stomatological Hospital, Capital Medical University
Other Study IDs: CMUSH-IRB-KJ-PJ-2020-10; Z191100006619042 (Other Grant/Funding Number: Beijing Municipal Science and Technology Commission)
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Oral Leukoplakia; Oral Cancer
Keywords: Oral cancer; Oral leukoplakia; Exosome; miR-185; Diagnosis; Prognosis
MeSH Terms: conditions — Leukoplakia, Oral; Mouth Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Saliva and plasma samples will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Detect the expression level of miR-185 in salivary and plasma exosomes. — Participants were instructed to refrain from eating, drinking, brushing their teeth, rinsing their mouth, or taking medications for one hour before saliva collection. They were then asked to bend over, lower their head, open their mouth, and allow saliva to flow naturally without chewing or spitting. Using a specialized container, 2 mL of unstimulated saliva was collected.
  Participants fasted overnight before blood collection. Researchers used plasma tubes containing anticoagulant (EDTA) to obtain venous blood (4-5 mL) from the participants' upper arm. Subsequently, the blood was gently inverted to ensure optimal contact with the anticoagulant before centrifugation at 2000 rpm and 4°C for 10 minutes. Following centrifugation, the supernatant was extracted.

SUMMARY:
The goal of this observational study is to test the expression levels of salivary and plasma exosomal miR-185 in patients with oral leukoplakia and oral squamous cell carcinoma. The main questions it aims to answer are:

* Is it possible to identify the cancer risk of oral leukoplakia in its early stages by detecting salivary and plasma exosomal miR-185?
* Is it possible to monitor the cancer risk of oral leukoplakia and the prognosis of oral cancer using salivary exosomal miR-185?

Participants will be asked to:

* Cooperate with the investigators in completing the oral examination.
* Take saliva and plasma before the biopsy surgery.
* Perform the biopsy surgery following the usual diagnostic procedures.
* Attend regular follow-up appointments (every 3 months) for the duration of the study.

DETAILED DESCRIPTION:
The first part of the study is a cross-sectional study in which the investigators will detect the expression level of salivary exosomal miR-185 in the participants at a single time point. The second part of the study is a prospective cohort study, in which the investigators will conduct regular follow-ups on the participants enrolled in the first part.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 30~80 years.
* Clinical diagnosis consistent with oral leukoplakia and oral cancer.
* Individuals with local stimulating factors correlated with oral lesions (including residual roots, residual crowns, poor oral restorations, cheek biting, and tongue biting habits).
* Oral lesions not subjected to any treatment, including laser, photodynamic therapy, radiotherapy, and chemotherapy.

Exclusion Criteria:

* Pathological diagnosis of another disease rather than oral leukoplakia or squamous cell carcinoma.
* Females who were pregnant or breastfeeding.
* Individuals who had malignancy, severe and precariously controlled diabetes mellitus, episodes of cardiovascular disease, hepatic or renal dysfunction, respiratory disease, hematologic disease, or immune abnormalities in the past year.
* Individuals with a psychiatric disorder.
* Other conditions deemed inappropriate for study participation by the researchers.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were from the Department of Stomatology, Beijing Stomatological Hospital, Capital Medical University, Beijing, China.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The expression level of miR-185 in salivary exosomes | Baseline, pre-biopsy surgery.
  Exosomes were isolated from saliva using ultracentrifugation, and total RNA from the exosomes was extracted using TRIzol reagent. Subsequently, the expression level of miR-185 was detected by RT-qPCR.
The expression level of miR-185 in plasma exosomes | Baseline, pre-biopsy surgery.
  Exosomes were isolated from plasma using ultracentrifugation, and total RNA from the exosomes was extracted using TRIzol reagent. Subsequently, the expression level of miR-185 was detected by RT-qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Guan, Ph.D., Study Director — Beijing Stomatological Hospital, Capital Medical University
Locations (1):
- Beijing Stomatological Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data on participants' gender, age, disease duration, lesion characteristics (location and size), tobacco, alcohol and betel nut consumption habits, histopathologic diagnosis, and miR-185 levels in saliva and plasma exosomes will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 years after publication of all results.
Access Criteria: Share data in a standardized format adhering to unified standards. The data should be comprehensive, trustworthy, traceable to the source, timely, and gathered and processed using consistent methods. Furthermore, anonymity of participants' identity information is required.
  Applicants seeking permission to access the data must clearly specify the intended purpose of use. Access to the data will only be granted to authorized individuals who have executed a data use agreement with the investigators. Any unauthorized sharing of data or use of the data for commercial purposes is strictly forbidden.
  Project Director Xiaobing Guan will be responsible for reviewing data access requests.
URL: http://www.medresman.org.cn

REFERENCES:
- [Background] Jing R, Chen W, Wang H, Ju S, Cong H, Sun B, Jin Q, Chu S, Xu L, Cui M. Plasma miR-185 is decreased in patients with esophageal squamous cell carcinoma and might suppress tumor migration and invasion by targeting RAGE. Am J Physiol Gastrointest Liver Physiol. 2015 Nov 1;309(9):G719-29. doi: 10.1152/ajpgi.00078.2015. Epub 2015 Aug 27. PMID 26316588
- [Background] Liu J, Han Y, Liu X, Wei S. Serum miR-185 Is a Diagnostic and Prognostic Biomarker for Non-Small Cell Lung Cancer. Technol Cancer Res Treat. 2020 Jan-Dec;19:1533033820973276. doi: 10.1177/1533033820973276. PMID 33251978
- [Background] Zhang W, Sun Z, Su L, Wang F, Jiang Y, Yu D, Zhang F, Sun Z, Liang W. miRNA-185 serves as a prognostic factor and suppresses migration and invasion through Wnt1 in colon cancer. Eur J Pharmacol. 2018 Apr 15;825:75-84. doi: 10.1016/j.ejphar.2018.02.019. Epub 2018 Feb 15. PMID 29454608
- [Background] Zhong WQ, Ren JG, Xiong XP, Man QW, Zhang W, Gao L, Li C, Liu B, Sun ZJ, Jia J, Zhang WF, Zhao YF, Chen G. Increased salivary microvesicles are associated with the prognosis of patients with oral squamous cell carcinoma. J Cell Mol Med. 2019 Jun;23(6):4054-4062. doi: 10.1111/jcmm.14291. Epub 2019 Mar 25. PMID 30907490
- [Background] Nieuwland R, Siljander PR. A beginner's guide to study extracellular vesicles in human blood plasma and serum. J Extracell Vesicles. 2024 Jan;13(1):e12400. doi: 10.1002/jev2.12400. PMID 38193375
- [Background] Witwer KW, Buzas EI, Bemis LT, Bora A, Lasser C, Lotvall J, Nolte-'t Hoen EN, Piper MG, Sivaraman S, Skog J, Thery C, Wauben MH, Hochberg F. Standardization of sample collection, isolation and analysis methods in extracellular vesicle research. J Extracell Vesicles. 2013 May 27;2. doi: 10.3402/jev.v2i0.20360. eCollection 2013. PMID 24009894
- [Background] Coumans FAW, Brisson AR, Buzas EI, Dignat-George F, Drees EEE, El-Andaloussi S, Emanueli C, Gasecka A, Hendrix A, Hill AF, Lacroix R, Lee Y, van Leeuwen TG, Mackman N, Mager I, Nolan JP, van der Pol E, Pegtel DM, Sahoo S, Siljander PRM, Sturk G, de Wever O, Nieuwland R. Methodological Guidelines to Study Extracellular Vesicles. Circ Res. 2017 May 12;120(10):1632-1648. doi: 10.1161/CIRCRESAHA.117.309417. PMID 28495994
- [Background] Vasconcelos MH, Caires HR, Abols A, Xavier CPR, Line A. Extracellular vesicles as a novel source of biomarkers in liquid biopsies for monitoring cancer progression and drug resistance. Drug Resist Updat. 2019 Dec;47:100647. doi: 10.1016/j.drup.2019.100647. Epub 2019 Oct 15. PMID 31704541
- [Background] Jeppesen DK, Fenix AM, Franklin JL, Higginbotham JN, Zhang Q, Zimmerman LJ, Liebler DC, Ping J, Liu Q, Evans R, Fissell WH, Patton JG, Rome LH, Burnette DT, Coffey RJ. Reassessment of Exosome Composition. Cell. 2019 Apr 4;177(2):428-445.e18. doi: 10.1016/j.cell.2019.02.029. PMID 30951670
- [Background] Vu LT, Gong J, Pham TT, Kim Y, Le MTN. microRNA exchange via extracellular vesicles in cancer. Cell Prolif. 2020 Nov;53(11):e12877. doi: 10.1111/cpr.12877. Epub 2020 Oct 6. PMID 33169503
- [Background] Li B, Cao Y, Sun M, Feng H. Expression, regulation, and function of exosome-derived miRNAs in cancer progression and therapy. FASEB J. 2021 Oct;35(10):e21916. doi: 10.1096/fj.202100294RR. PMID 34510546
- [Background] Lu TX, Rothenberg ME. MicroRNA. J Allergy Clin Immunol. 2018 Apr;141(4):1202-1207. doi: 10.1016/j.jaci.2017.08.034. Epub 2017 Oct 23. PMID 29074454
- [Background] Mathieu M, Martin-Jaular L, Lavieu G, Thery C. Specificities of secretion and uptake of exosomes and other extracellular vesicles for cell-to-cell communication. Nat Cell Biol. 2019 Jan;21(1):9-17. doi: 10.1038/s41556-018-0250-9. Epub 2019 Jan 2. PMID 30602770
- [Background] Wang L, Yin P, Wang J, Wang Y, Sun Z, Zhou Y, Guan X. Delivery of mesenchymal stem cells-derived extracellular vesicles with enriched miR-185 inhibits progression of OPMD. Artif Cells Nanomed Biotechnol. 2019 Dec;47(1):2481-2491. doi: 10.1080/21691401.2019.1623232. PMID 31219352